CLINICAL TRIAL: NCT07233135
Title: The Effect of Different Materials on Students' Learning Satisfaction and Self-Confidence in Episiotomy Education: A Randomized Quasi-Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Melek Şen Aytekin, Research Assistant Doctor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GaziosmanpasaU-EBE-MŞA-03
Record Dates: First submitted 2025-10-02; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Education
Keywords: midwifery; education; episiotomy; simulation; chichen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Episiotomy Simulation Model (Experimental): This group received online episiotomy repair training as part of the Normal Birth and Postpartum Term course. The training was delivered as two 60-minute lessons using PowerPoint presentations. The training included a video of episiotomy repair prepared by the researchers. Following the training, the first researcher demonstrated episiotomy repair on a simulation model in a laboratory setting. The students then performed the procedure on chicken breasts.
  Interventions: Other: Episiotomy Simulation Model
- Chicken Breast Group (Experimental): This group received online episiotomy repair training as part of the Normal Birth and Postpartum Term course. The training was delivered as two 60-minute lessons using PowerPoint presentations. The training included watching an episiotomy repair video prepared by the researchers. Following the training, the first researcher demonstrated episiotomy repair on a chicken breast in a laboratory setting. The students then performed the procedure on the chicken breast.
  Interventions: Other: Chicken Breast Group

INTERVENTIONS:
Other: Chicken Breast Group — Chicken breast is dead animal tissue that can be used to practice repairing lacerations or episiotomies following vaginal delivery. The chicken breast was used. The impact of working with this model on students' satisfaction and self-confidence was investigated, and its suitability for simulation was evaluated.
  Arms: Chicken Breast Group
Other: Episiotomy Simulation Model — The Episiotomy Simulation Model provides a realistic tool for practicing the care and repair of lacerations or apisiotomies following vaginal delivery. The impact of working with this model on students' satisfaction and self-confidence was investigated, and the suitability of the simulation was evaluated.
  Arms: Episiotomy Simulation Model

SUMMARY:
As part of this research, episiotomy training for third-year midwifery students was transformed into an online video-assisted process due to the pandemic. The aim of the training was to determine the impact of episiotomy repair practice with different materials in a laboratory setting on students' satisfaction and self-confidence and to evaluate the suitability of the simulation design.

DETAILED DESCRIPTION:
This study was conducted to determine the effects of episiotomy repair training on learning satisfaction and self-confidence using different materials and to determine the suitability of the materials for learning.

The standard training was provided to midwifery students online via video support due to the pandemic. Following a power analysis, a total of 52 students were planned to be enrolled, 26 in each group. However, due to student withdrawals or exclusions during the study, which occurred with varying degrees of difficulty, the study was completed with a total of 43 students.

The online standard training was delivered to all students as two 60-minute lessons using a PowerPoint presentation. Following the training, the researchers watched an episiotomy skills training video, created using a mock-up model. Pre-tests were completed after the standard training period was completed. A personal information form and the Student Satisfaction with Learning and Self-Confidence Scale were used in the pre-tests.

The students were randomly assigned to two treatment groups: "Chicken Breast" and "Episiotomy Simulation Model." The first researcher demonstrated episiotomy repair on the material according to their group. In accordance with the training provided, students performed episiotomy repairs using materials in their laboratory group. After completing the exercises, students were administered post-tests. In these post-tests, students completed the Student Satisfaction and Self-Confidence in Learning Scale and the Simulation Design Scale.

ELIGIBILITY:
Inclusion Criteria:

* Third-year midwifery students who volunteered to participate in the study,
* were taking a course on normal birth and the postpartum period for the first time, had no experience with episiotomy repair, and had not previously observed an episiotomy repair procedure, were included in the study.

Exclusion Criteria:

* Students who were absent on the day the episiotomy topic was taught.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Simulation Design Scale | Used 5 minutes after the students performed the episiotomy repair, depending on their group.
  The scale consists of 20 items and 5 subscales. The Goals and Information subscale consists of 5 items, the Support subscale consists of 4 items, the Problem Solving subscale consists of 5 items, the Feedback/Guided Reflection subscale consists of 4 items, and the Degree of Realism subscale consists of 2 items. The total Cronbach's alpha value for the scale is 0.90. The scale consists of two sections: one for evaluating the simulation model and one for assessing the importance of the simulation design. The first section is rated as "strongly disagree with the statement," "disagree with the statement," "undecided," "agree with the statement," "strongly agree with the statement," and "not applicable." The second section is rated as "not important," "somewhat important," "undecided," "important," and "very important." Scale scores are obtained by dividing the total and subscale scores by the number of items
Student Satisfaction-Self-Confidence in Learning Scale | It was used 5 minutes after completing standard training. It was also used 5 minutes after the students performed the episiotomy repair, depending on their group.
  The scale was developed by Jeffries and Rizzolo (2006) and consists of two subscales: satisfaction with current learning (5 items) and self-confidence in learning (8 items). The scale does not contain any reverse items. Validity and reliability for the Turkish version were conducted by Ünver et al. (2017). The Turkish version of the scale consists of 13 items. It is a five-point Likert-type scale (values range from strongly disagree (1) to strongly agree (5)). The total scale score is obtained by dividing the subscale score by the number of items. A high total score indicates that student satisfaction and self-confidence in learning are high.

SECONDARY OUTCOMES:
Personal Information Form | Used 5 minutes after completing standard training.
  This form was developed by researchers to determine the demographic characteristics of students, based on literature. It consists of questions that include introductory information about students, such as their age, previous education, reasons for choosing their profession, and their level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No